CLINICAL TRIAL: NCT05590650
Title: A Pilot Study of Additional Chinese Formula for Concurrent Chemoradiotherapy in Oral Cavity Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CMUH106-REC3-149
Record Dates: First submitted 2022-10-16; First posted 2022-10-21 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Head and Neck Neoplasm; Chemoradiotherapy
Keywords: Head and Neck Neoplasms;; Chemoradiotherapy; Complementary Therapies; Medicine, Chinese Traditional
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SZKJT group (Experimental): Patients who meet the inclusion criteria and agree to receive concomitant treatment with SZKJT.
  Interventions: Drug: SZKJT(San-Zhong-Kui-Jian-Tang)

INTERVENTIONS:
Drug: SZKJT(San-Zhong-Kui-Jian-Tang) — The SZKJT samples were made and packed by Kaiser Pharmaceutical Co. Ltd. with lot number of 2019023247.
  Other Names: Product from Kaiser Pharmaceutical Co. Ltd.

SUMMARY:
The goal of this clinical trial is to learn about the clinical efficacy of San-Zhong-Kui-Jian-Tang (SZKJT), a formula of Chinese medicine in head and neck cancer patients receiving concurrent chemoradiotherapy (CCRT) treatments. The main questions it aims to answer are:

* Can SZKJT improve the completion rate of CCRT?
* Can SZKJT reduce the adverse effects of CCRT?
* How SZKJT affect the quality of life in the patients receiving CCRT
* How about the safety of using SZKJT in the patients receiving CCRT

Participants will be asked to:

* take SZKJT for 9 weeks during the whole CCRT course
* take questionnaires of quality of life

DETAILED DESCRIPTION:
San-Zhong-Kui-Jian-Tang (SZKJT) is originated from the Secret Treasure of the Orchid Chamber written by Gao Li (AC1180 - 1251). SZKJT contains 16 herbs to treat abnormal swelling or nodules. In the theory of Chinese medicine, SZKJT can clear heat and resolve toxin, which leads to disperse swelling and binds in nodules.

The purpose of this study is to explore the clinical efficacy and safety of SZKJT in improving the completion rate of concurrent chemoradiotherapy (CCRT) in patients with head and neck cancer, and to evaluate the prevention and treatment effects of SZKJT on the side effects of chemoradiotherapy, as well as the improvement of quality of life.

The primary endpoint of the study is the completion rate of CCRT under SZKJT treatment. The secondary endpoints are adverse effects of CTCAE, body constitution questionnaire (BCQ) and the EORTC core quality of life questionnaire (QLQ-C30). Liver and kidney functions are considered as well for adverse effects of SZKJT. We hypothesized that additional SZKJT with CCRT might improve completion rate of CCRT and reduce severity of adverse effects of CCRT.

ELIGIBILITY:
Inclusion Criteria:

* aged from 20- to 65-year-old;
* firstly diagnosed as head and neck cancer with stage II, III or IV;
* adjuvant therapy with chemotherapy of Cisplatin or combined with radiotherapy after surgery;
* or chemotherapy of Cisplatin for those without surgery;
* wiliness to sign inform consent.

Exclusion Criteria:

* pregnancy;
* non-Squamous-cell carcinoma;
* secondary cancer or Carcinoma in situ in 5 years;
* any evidence of metastasis;
* abnormality of liver, kidney or bone marrow functions before treatments;
* unstable vital signs;
* episode of acute infection;
* unclear consciousness for inform consent;
* receiving other herbal, complementary or acupuncture therapy.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-07-07 (Actual); Primary Completion 2020-06-14 (Actual); Study Completion 2020-12-25 (Actual)

PRIMARY OUTCOMES:
The completion rate | We will do an assessment at the seventh week of CCRT. Patients who had completed a seven-week course of treatment and had a cumulative dose of cisplatin greater than 200 mg per m2 will be considered the completion group.
  We counted the percentage rate of those who achieved and did not reach the CCRT course.

SECONDARY OUTCOMES:
The adverse effects | The assessment is performed at the eighth week.
  We apply Common Terminology Criteria for Adverse Events (CTCAE) to assess the adverse effects of CCRT.
The change in Quality of Life | The questionnaire is assessed at the baseline and the eighth week.
  We assess the patients' quality of life by using the European Organisation for Research and Treatment of Cancer (EORTC) quality-of-life questionnaire QLQ-C30.
The Change of Constitutions of traditional Chinese medicine | The questionnaire is assessed at the baseline and the eighth week.
  We assess the patients' constitutions of traditional Chinese medicine by using Body Constitution Questionnaire (BCQ).
The change of liver function | The lab data of biochemistry analysis is collected at the baseline and the eighth week.
  We monitor the liver function of the patients by blood chemistry analysis. The levels of Alanine transaminase (ALT) and Aspartate transaminase (AST) are recorded as units per liter.
The change of renal function | The lab data of biochemistry analysis is collected at the baseline and the eighth week.
  We monitor the renal function of the patients by blood chemistry analysis. The levels of blood urine nitrogen (mg/dL) and creatinine (mg/dL) are recorded. Glomerular filtration rate (GFR) is estimated by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) Creatinine Equation (2021).

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Yu Lien, Ph.D, Principal Investigator — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bernier J, Domenge C, Ozsahin M, Matuszewska K, Lefebvre JL, Greiner RH, Giralt J, Maingon P, Rolland F, Bolla M, Cognetti F, Bourhis J, Kirkpatrick A, van Glabbeke M; European Organization for Research and Treatment of Cancer Trial 22931. Postoperative irradiation with or without concomitant chemotherapy for locally advanced head and neck cancer. N Engl J Med. 2004 May 6;350(19):1945-52. doi: 10.1056/NEJMoa032641. PMID 15128894
- [Background] Cooper JS, Pajak TF, Forastiere AA, Jacobs J, Campbell BH, Saxman SB, Kish JA, Kim HE, Cmelak AJ, Rotman M, Machtay M, Ensley JF, Chao KS, Schultz CJ, Lee N, Fu KK; Radiation Therapy Oncology Group 9501/Intergroup. Postoperative concurrent radiotherapy and chemotherapy for high-risk squamous-cell carcinoma of the head and neck. N Engl J Med. 2004 May 6;350(19):1937-44. doi: 10.1056/NEJMoa032646. PMID 15128893
- [Background] Bernier J, Cooper JS, Pajak TF, van Glabbeke M, Bourhis J, Forastiere A, Ozsahin EM, Jacobs JR, Jassem J, Ang KK, Lefebvre JL. Defining risk levels in locally advanced head and neck cancers: a comparative analysis of concurrent postoperative radiation plus chemotherapy trials of the EORTC (#22931) and RTOG (# 9501). Head Neck. 2005 Oct;27(10):843-50. doi: 10.1002/hed.20279. PMID 16161069
- [Background] Cooper JS, Zhang Q, Pajak TF, Forastiere AA, Jacobs J, Saxman SB, Kish JA, Kim HE, Cmelak AJ, Rotman M, Lustig R, Ensley JF, Thorstad W, Schultz CJ, Yom SS, Ang KK. Long-term follow-up of the RTOG 9501/intergroup phase III trial: postoperative concurrent radiation therapy and chemotherapy in high-risk squamous cell carcinoma of the head and neck. Int J Radiat Oncol Biol Phys. 2012 Dec 1;84(5):1198-205. doi: 10.1016/j.ijrobp.2012.05.008. Epub 2012 Jun 30. PMID 22749632
- [Background] Forastiere AA, Goepfert H, Maor M, Pajak TF, Weber R, Morrison W, Glisson B, Trotti A, Ridge JA, Chao C, Peters G, Lee DJ, Leaf A, Ensley J, Cooper J. Concurrent chemotherapy and radiotherapy for organ preservation in advanced laryngeal cancer. N Engl J Med. 2003 Nov 27;349(22):2091-8. doi: 10.1056/NEJMoa031317. PMID 14645636
- [Background] Adelstein DJ, Li Y, Adams GL, Wagner H Jr, Kish JA, Ensley JF, Schuller DE, Forastiere AA. An intergroup phase III comparison of standard radiation therapy and two schedules of concurrent chemoradiotherapy in patients with unresectable squamous cell head and neck cancer. J Clin Oncol. 2003 Jan 1;21(1):92-8. doi: 10.1200/JCO.2003.01.008. PMID 12506176
- [Background] Trotti A, Bellm LA, Epstein JB, Frame D, Fuchs HJ, Gwede CK, Komaroff E, Nalysnyk L, Zilberberg MD. Mucositis incidence, severity and associated outcomes in patients with head and neck cancer receiving radiotherapy with or without chemotherapy: a systematic literature review. Radiother Oncol. 2003 Mar;66(3):253-62. doi: 10.1016/s0167-8140(02)00404-8. PMID 12742264
- [Background] Russo G, Haddad R, Posner M, Machtay M. Radiation treatment breaks and ulcerative mucositis in head and neck cancer. Oncologist. 2008 Aug;13(8):886-98. doi: 10.1634/theoncologist.2008-0024. Epub 2008 Aug 13. PMID 18701763
- [Background] Robertson AG, Robertson C, Perone C, Clarke K, Dewar J, Elia MH, Hurman D, MacDougall RH, Yosef HM. Effect of gap length and position on results of treatment of cancer of the larynx in Scotland by radiotherapy: a linear quadratic analysis. Radiother Oncol. 1998 Aug;48(2):165-73. doi: 10.1016/s0167-8140(98)00038-3. PMID 9783888
- [Background] Robertson C, Robertson AG, Hendry JH, Roberts SA, Slevin NJ, Duncan WB, MacDougall RH, Kerr GR, O'Sullivan B, Keane TJ. Similar decreases in local tumor control are calculated for treatment protraction and for interruptions in the radiotherapy of carcinoma of the larynx in four centers. Int J Radiat Oncol Biol Phys. 1998 Jan 15;40(2):319-29. doi: 10.1016/s0360-3016(97)00716-5. PMID 9457816
- [Background] Groome PA, O'Sullivan B, Mackillop WJ, Jackson LD, Schulze K, Irish JC, Warde PR, Schneider KM, Mackenzie RG, Hodson DI, Hammond JA, Gulavita SP, Eapen LJ, Dixon PF, Bissett RJ. Compromised local control due to treatment interruptions and late treatment breaks in early glottic cancer: Population-based outcomes study supporting need for intensified treatment schedules. Int J Radiat Oncol Biol Phys. 2006 Mar 15;64(4):1002-12. doi: 10.1016/j.ijrobp.2005.10.010. Epub 2006 Jan 18. PMID 16414205
- [Background] Herrmann T, Jakubek A, Trott KR. The importance of the timing of a gap in radiotherapy of squamous cell carcinomas of the head and neck. Strahlenther Onkol. 1994 Sep;170(9):545-9. PMID 7940126
- [Background] Thomas K, Martin T, Gao A, Ahn C, Wilhelm H, Schwartz DL. Interruptions of Head and Neck Radiotherapy Across Insured and Indigent Patient Populations. J Oncol Pract. 2017 Apr;13(4):e319-e328. doi: 10.1200/JOP.2016.017863. Epub 2017 Mar 7. PMID 28267393
- [Background] Suwinski R, Sowa A, Rutkowski T, Wydmanski J, Tarnawski R, Maciejewski B. Time factor in postoperative radiotherapy: a multivariate locoregional control analysis in 868 patients. Int J Radiat Oncol Biol Phys. 2003 Jun 1;56(2):399-412. doi: 10.1016/s0360-3016(02)04469-3. PMID 12738315
- [Derived] Tang HT, Ou SC, Chu CL, Lee AL, Lin HJ, Lin YC, Wang YC, Yang SN, Lien MY. Chinese Herbal Medicine for Concurrent Chemoradiation-Induced Adverse Events in Head and Neck Cancer Patients: A Prospective Feasibility Study. Integr Cancer Ther. 2025 Jan-Dec;24:15347354251326946. doi: 10.1177/15347354251326946. Epub 2025 Mar 24. PMID 40123292